CLINICAL TRIAL: NCT05583149
Title: A Phase 2 Study of Acalabrutinib in Combination With Lisocabtagene Maraleucel in Relapsed/Refractory Aggressive B-cell Lymphomas
Brief Title: Acalabrutinib + Liso-Cel In R/R Aggressive B-Cell Lymphomas
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Patrick C. Johnson, MD (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Patrick C. Johnson, MD, Sponsor Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 21-422
Record Dates: First submitted 2022-10-13; First posted 2022-10-17 (Actual); Results first posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Refractory Aggressive B-cell Lymphomas; Refractory B-Cell Non-Hodgkin Lymphoma; Aggressive B-cell NHL; Diffuse Large B-cell Lymphoma (DLBCL); De Novo or Transformed Indolent B-cell Lymphoma; DLBCL, Nos Genetic Subtypes; T Cell/Histiocyte-rich Large B-cell Lymphoma; EBV-Positive DLBCL, Nos; Primary Mediastinal [Thymic] Large B-cell Lymphoma (PMBCL); High-Grade B-Cell Lymphoma, Nos; C-MYC/BCL6 Double-Hit High-Grade B-Cell Lymphoma; Grade 3b Follicular Lymphoma; C-MYC/BCL2 Double-Hit High-Grade B-Cell Lymphoma
Keywords: Refractory aggressive B-cell lymphomas; Refractory B-Cell Non-Hodgkin Lymphoma; Aggressive B-cell NHL; Diffuse Large B-cell Lymphoma (DLBCL); De novo or transformed indolent B-cell lymphoma; DLBCL, nos Genetic Subtypes; T cell/histiocyte-rich large B-cell lymphoma; EBV-Positive DLBCL, nos; Primary mediastinal [thymic] large B-cell lymphoma (PMBCL); High-Grade B-Cell Lymphoma, nos; C-MYC/BCL6 Double-Hit High-Grade B-Cell Lymphoma; Grade 3b Follicular Lymphoma; C-MYC/BCL2 Double-Hit High-Grade B-Cell Lymphoma
MeSH Terms: conditions — Lymphoma, B-Cell; Lymphoma, Large B-Cell, Diffuse; Pyloric Stenosis, Hypertrophic | interventions — acalabrutinib; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ACALABRUTINIB and LISOCABTAGENE MARALEUCEL (Experimental): The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits, as tolerated for one year
  * Liso-cel
  * Acalabrutinib
  Interventions: Drug: ACALABRUTINIB; Drug: LISOCABTAGENE MARALEUCEL; Drug: Lymphodepleting chemotherapy

INTERVENTIONS:
Drug: ACALABRUTINIB — Oral, twice daily, timing and dosage per protocol
  Other Names: Calquence
Drug: LISOCABTAGENE MARALEUCEL — via IV timings and dosage per protocol
  Other Names: Breyanzi
Drug: Lymphodepleting chemotherapy — lymphodepleting chemotherapy with cyclophosphamide and fludarabine once a day for 3 days via IV about 2-4 hours. This will occur only once prior to lisocabtagene maraleucel infusion.
  Other Names: cyclophosphamide and fludarabine

SUMMARY:
This research is being done to assess the effectiveness and safety of acalabrutinib combined with lisocabtagene maraleucel (liso-cel) for people with relapsed/refractory aggressive B-cell lymphoma.

This research study involves the study drug acalabrutinib in combination with lisocabtagene maraleuce

DETAILED DESCRIPTION:
This research study involves the study drug acalabrutinib in combination with lisocabtagene maraleucel.

The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits.

- Participants will receive one infusion of liso-cel and will receive acalabrutinib capsules twice daily as long as treatment is tolerated and disease does not worsen (disease progression) for up to one year.

Participants will be followed by clinical visits for up to 5 years and the medical record will be monitored for up to 15 years.

It is expected that about 27 people will take part in this research study.

This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

The U.S. Food and Drug Administration (FDA) has not approved acalabrutinib for this specific disease, but it has been approved for other uses.

The U.S. FDA has approved lisocabtagene maraleucel for this specific disease.

AstraZeneca, a pharmaceutical company, is supporting this research study by providing funding for the research study and supplying acalabrutinib.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients ≥18 years with histologically confirmed aggressive B-cell NHL including diffuse large B-cell lymphoma (DLBCL), either de novo or transformed from any indolent B-cell lymphoma, and including DLBCL NOS, T cell/histiocyte-rich large B-cell lymphoma, Epstein-Barr virus [EBV] positive DLBCL NOS, primary mediastinal [thymic] large B-cell lymphoma (PMBCL), high grade B-cell lymphoma NOS, or high grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangements [double/triple hit lymphoma (DHL/THL)]; and grade 3B follicular lymphoma. Patients with primary CNS lymphoma are not eligible. Patients with secondary CNS involvement by lymphoma are eligible if they otherwise meet all eligibility criteria.
* Relapsed or refractory to at least 2 prior lines of systemic lymphoma therapy. Previous therapy must have included a CD20-targeted agent and an anthracycline or alkylating agent.
* PET-positive measurable disease
* ECOG Performance status 0-2
* Estimated creatinine clearance of ≥30 mL/min, calculated using the Cockcroft and Gault equation (if male, [140Age] x Mass [kg] / [72 x creatinine g/dL];multiply by 0.85 if female)
* Alanine Aminotransferase (ALT) <= 2.5 times the ULN
* Bilirubin <= 2 x ULN (or <= 3.0 mg/dL for patients with Gilbert-Meulengracht syndrome or lymphomatous involvement of the liver)
* Hemodynamically stable and Left Ventricle Ejection Fraction (LVEF) >= 40% confirmed by echocardiogram or Multigated Radionuclide Angiography (MUGA)
* For subjects with atrial fibrillation, atrial fibrillation must be controlled and asymptomatic
* Absolute neutrophil count (ANC) >= 1000/mm3
* Platelets >= 50,000/mm3
* Adequate pulmonary function, defined as <= CTCAE Grade 1 dyspnea and SaO2 > 91% on room air
* Adequate vascular access for leukapheresis procedure (either peripheral line or surgically-placed line)
* Woman of childbearing potential (WOCBP) who are sexually active must use highly effective methods of contraception during treatment and for 2 days after the last dose of acalabrutinib.
* Willing and able to participate in all required evaluations and procedures in this study protocol.
* Ability to understand the purpose and risks of the study and provide signed and dated informed consent and authorization to use protected health information.

Exclusion Criteria:

* Another active malignancy which requires concurrent cancer-directed therapy
* Previous treatment with gene therapy product or adoptive T cell therapy
* Allogeneic stem cell transplant within 90 days of leukapheresis
* Active acute or chronic GVHD
* HIV infection
* Serologic status reflecting active hepatitis B or C infection

  * Subjects who are hepatitis B core antibody (anti-HBc) positive and who are hepatitis B surface antigen (HBsAg) negative will need to have a negative PCR result before enrollment and must be willing to undergo DNA PCR testing during the study. Those who are HbsAg-positive or hepatitis B PCR positive will be excluded.
  * Subjects who are hepatitis C antibody positive will need to have a negative PCR result before enrollment. Those who are hepatitis C PCR positive will be excluded.
* Uncontrolled infection
* Clinically relevant CNS pathology
* History of cardiovascular conditions within the past 6 months, including class III or IV heart failure as defined by New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or clinically significant arrhythmias: Participants with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, participants should be class 2B or better.
* Autoimmune disease requiring chronic systemic corticosteroids at a dose of greater than 10 mg of prednisone daily or an equivalent dose of another corticosteroid
* Treatment with alemtuzumab within 6 months leukapheresis or fludarabine or cladribine within 3 months of leukapheresis
* Therapeutic anticoagulation
* Bleeding diathesis
* Has difficulty with or is unable to swallow oral medication, or has significant gastrointestinal disease that would limit absorption of oral medication.
* Known history of hypersensitivity or anaphylaxis to study drug(s) including active product or excipient components.
* Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening.
* Requires treatment with a strong cytochrome P450 3A4 (CYP3A4) inhibitor/inducer.
* Prothrombin time (PT)/INR or aPTT (in the absence of lupus anticoagulant) >2x ULN.
* Requires treatment with proton pump inhibitors (eg, omeprazole, esomeprazole, lansoprazole, dexlansoprazole, rabeprazole, or pantoprazole). Note: Subjects receiving proton pump inhibitors who switch to H2-receptor antagonists or antacids are eligible for enrollment to this study.
* History of significant cerebrovascular disease/event, including stroke or intracranial hemorrhage, within 6 months before the first dose of study drug.
* Major surgical procedure within 28 days of first dose of study drug. Note: If a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
* Breastfeeding or pregnant: Pregnant women are excluded from this study because acalabrutinib is an agent with the potential for teratogenic or abortifacient effects.

Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with acalabrutinib, breastfeeding should be discontinued if the mother is treated with acalabrutinib.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-11-23 (Actual); Study Completion 2029-03-01 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Connor Johnson, MD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth-Israel Deaconess Medical Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | ACALABRUTINIB and LISOCABTAGENE MARALEUCEL
Started | 28
Completed | 26
Not Completed | 2
Not completed — Development of concurrent medical condition that interferes with trial participation | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Groups:
- ACALABRUTINIB and LISOCABTAGENE MARALEUCEL: The research study procedures include screening for eligibility and study treatment including evaluations and follow up visits, as tolerated for one year
  * Liso-cel
  * Acalabrutinib
  ACALABRUTINIB: Oral, twice daily, timing and dosage per protocol
  LISOCABTAGENE MARALEUCEL: via IV timings and dosage per protocol
  Lymphodepleting chemotherapy: lymphodepleting chemotherapy with cyclophosphamide and fludarabine once a day for 3 days via IV about 2-4 hours. This will occur only once prior to lisocabtagene maraleucel infusion.
Arm/Group | ACALABRUTINIB and LISOCABTAGENE MARALEUCEL
Number analyzed (Participants) | 28
Age, Continuous [Median (Full Range); unit: years] | 70 [28 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 16
  More than one race | 1
  Unknown or Not Reported | 6

OUTCOME MEASURES:

1. Primary Outcome: Complete Response Rate (CRR)
Description: The CRR is defined as the percentage of subjects achieving an objective response of complete response (CR) according to the Lugano Classification (Chesson et al., 2014), prior to start of another non-study anticancer therapy. CR is defined as a complete metabolic and radiologic response (Lugano score 1-3, target nodes/nodal masses must regress to ≤ 1.5 cm in longest diameter.)
Time Frame: 1 year 8 months
Measure: Count of Participants; unit: Participants
Arm/Group | ACALABRUTINIB and LISOCABTAGENE MARALEUCEL
Number analyzed (Participants) | 27
Participants | 22

2. Secondary Outcome: Overall Response Rate
Time Frame: 3 Months
Reporting Status: Not Posted

3. Secondary Outcome: Overall Response Rate
Time Frame: 6 Months
Reporting Status: Not Posted

4. Secondary Outcome: Overall Response Rate
Time Frame: 12 Months
Reporting Status: Not Posted

5. Secondary Outcome: Progression Free Survival
Description: PFS will be summarized using Kaplan-Meier estimates.
Time Frame: as the time from registration to the earlier of progression or death due to any cause. Participants alive without disease progression are censored at date of last disease evaluation up to 15 years
Reporting Status: Not Posted

6. Secondary Outcome: Overall Survival
Description: OS will be summarized using Kaplan- Meier estimates.
Time Frame: defined as the time from registration to death due to any cause, or censored at date last known alive up to 15 years
Reporting Status: Not Posted

7. Secondary Outcome: Duration of Response
Description: The duration of overall response is measured from the time measurement criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented (taking as reference for progressive disease the smallest measurements recorded since the treatment started, or death due to any cause. Participants without events reported are censored at the last disease evaluation).DOR will be summarized using Kaplan-Meier estimates.
Time Frame: time from first response to disease progression or death up to 15 years
Reporting Status: Not Posted

8. Secondary Outcome: Event Free Survival
Description: Time to event outcomes will be estimated using Kaplan Meier method or cumulative incidence curves
Time Frame: from registration to death from any cause, disease progression, or starting a new anti-lymphoma therapy, whichever occurs first up to 15 years
Reporting Status: Not Posted

9. Secondary Outcome: Rates of Bridging Therapy
Description: Rates of bridging therapy defined as the percentage of participants requiring any lymphoma-directed therapy other than the investigational therapy in order to control the disease prior to liso-cel infusion. Reported with descriptive statistics
Time Frame: 1 years
Reporting Status: Not Posted

10. Secondary Outcome: FACT-G QOL
Description: Functional Assessment of Cancer Treatment-General (FACT-G). The FACT-G consists of four subscales assessing well-being across four domains. These self-reported measures possess strong psychometric properties and have been validated for patients with cancer
Time Frame: baseline, day -5 (+/- 3 days), day +7 (+/- 3 days), day +30 (+/- 7 days), day +90 (+/- 14 days), and day +180 (+/- 14 days) after liso-cel infusion
Reporting Status: Not Posted

11. Secondary Outcome: ICU Rates
Description: ICU admission rates defined as the percentage of participants with an ICU admission within 90 days of liso-cel infusion. Reported with descriptive statistics
Time Frame: up to 90 days
Reporting Status: Not Posted

12. Secondary Outcome: Re-hospitalization Rates
Description: All cause re-hospitalization rates defined as the percentage of participants who experience an unplanned hospitalization within 90 days of liso-cel infusion. Planned hospital admissions for a procedure or treatment will be excluded. Reported with descriptive statistics
Time Frame: up to 90 days
Reporting Status: Not Posted

13. Secondary Outcome: ER Visit Rates
Description: All cause ER visit rates defined as the percentage of participants who experience an unplanned ER visit within 90 days of liso-cel infusion.
  Planned ER visits/hospital admissions for a procedure or treatment will be excluded.
Time Frame: within 90 days
Reporting Status: Not Posted

14. Secondary Outcome: Length of Stay
Description: Length of stay (LOS) defined as the number of days a participant is hospitalized for liso-cel infusion.
Time Frame: 1 year
Reporting Status: Not Posted

15. Secondary Outcome: Rates of Acalabrutinib Discontinuation Due to Toxicity
Description: Rates of acalabrutinib discontinuation in participants due to acalabrutinib toxicity NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Time Frame: time of their first treatment up to 3 years
Reporting Status: Not Posted

16. Secondary Outcome: Number of Participants Treatment Related Adverse Event NCI CTCAE 5.0
Description: The descriptions and grading scales found in the revised NCI Common Terminology Criteria for Adverse Events (CTCAE) version 5.0
Time Frame: up to 3 Years
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All adverse events are reported from the start of acalabrutinib until 30 days after the last dose of study drug or at documented disease progression, whichever is longer. For patients without disease progression at 90 days after the last dose of study drug, only adverse events at least possibly related to study drug are reported through year 2 or disease progression, whichever occurs first (adverse events followed up to 24 months in a single patient as of November 2025.)
Arm/Group | ACALABRUTINIB and LISOCABTAGENE MARALEUCEL
All-Cause Mortality (participants affected / at risk) | 0/27
Serious Adverse Events (participants affected / at risk) | 7/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACALABRUTINIB and LISOCABTAGENE MARALEUCEL (N=27)
Alanine aminotransferase increased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Cytokine Release Syndrome (Investigations) | 1
Fever (General disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hypotension (Vascular disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Neck mass
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ACALABRUTINIB and LISOCABTAGENE MARALEUCEL (N=27)
Abdominal infection (Infections and infestations) | 1
Abdominal Pain (Gastrointestinal disorders) | 5
Agitation (Psychiatric disorders) | 1
Alanine aminotransferase increased (Investigations) | 5
Alkaline phosphatase increased (Investigations) | 2
Allergic reaction (Immune system disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 4
Alopecia (Skin and subcutaneous tissue disorders) | 2
Anemia (Blood and lymphatic system disorders) | 6
Anorexia (Metabolism and nutrition disorders) | 9
Anxiety (Psychiatric disorders) | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 5
Aspartate aminotransferase increased (Investigations) | 5
Atrial fibrillation (Cardiac disorders) | 4
Atrial flutter (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 9
Bacteremia (Infections and infestations) | 1
Bloating (Gastrointestinal disorders) | 3
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 4 — hypogammaglobulinemia
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1 — Bleeding (Peripherally Inserted Central Catheter site)
Blood antidiuretic hormone abnormal (Investigations) | 1
Blood bilirubin increased (Investigations) | 1
Blurred vision (Eye disorders) | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Bronchial infection (Infections and infestations) | 1
Bronchial stricture (Respiratory, thoracic and mediastinal disorders) | 1
Bruising (Injury, poisoning and procedural complications) | 5
Cataract (Eye disorders) | 1
Chills (General disorders) | 3
Chronic kidney disease (Renal and urinary disorders) | 1
Cognitive disturbance (Nervous system disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 15
Cough (Respiratory, thoracic and mediastinal disorders) | 13
Creatinine increased (Investigations) | 4
Cytokine release syndrome (Immune system disorders) | 16
Dehydration (Metabolism and nutrition disorders) | 15
Depression (Psychiatric disorders) | 3
Diarrhea (Gastrointestinal disorders) | 12
Dizziness (Nervous system disorders) | 14
Dry eye (Eye disorders) | 2
Dry mouth (Gastrointestinal disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Dysarthria (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 2
Dyspepsia (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 7
Dysuria (Renal and urinary disorders) | 2
Ear and labyrinth disorders - Other, specify (Ear and labyrinth disorders) | 1 — Hearing loss (left ear)
Edema face (General disorders) | 1
Edema limbs (General disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 2 — Subconjunctival Hemorrhage
Eye disorders - Other, specify (Eye disorders) | 1 — Vitreous detachment
Eye disorders - Other, specify (Eye disorders) | 1 — diplopia
Fall (Injury, poisoning and procedural complications) | 2
Fatigue (General disorders) | 23
Febrile neutropenia (Blood and lymphatic system disorders) | 8
Fecal incontinence (Gastrointestinal disorders) | 4
Fever (General disorders) | 10
Fibrinogen decreased (Investigations) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Flu like symptoms (General disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 9
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — abdominal cramping
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 1 — Diverticulitis
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Decreased oral intake
General disorders and administration site conditions - Other, specify (General disorders) | 1 — Chest Tightness
Glucose intolerance (Metabolism and nutrition disorders) | 1
Headache (Nervous system disorders) | 13
Hearing impaired (Ear and labyrinth disorders) | 1
Heart failure (Cardiac disorders) | 1
Hematoma (Vascular disorders) | 1
Hemorrhoids (Gastrointestinal disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 4
Dysphasia (Nervous system disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5
Hyperlipidemia (Metabolism and nutrition disorders) | 7
Hypertension (Vascular disorders) | 11
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypokalemia (Metabolism and nutrition disorders) | 8
Hypomagnesemia (Metabolism and nutrition disorders) | 7
Hyponatremia (Metabolism and nutrition disorders) | 7
Hypophosphatemia (Metabolism and nutrition disorders) | 8
Hypotension (Vascular disorders) | 12
Hypothermia (General disorders) | 3
Hypothyroidism (Endocrine disorders) | 2
Immune system disorders - Other, specify (Immune system disorders) | 1 — immune effector cell-associated haemophagocytic lymphohistiocytosis-like syndrome
Infections and infestations - Other, specify (Infections and infestations) | 6 — Covid-19
Infections and infestations - Other, specify (Infections and infestations) | 1 — Viral Infection
Infusion related reaction (Injury, poisoning and procedural complications) | 1
INR increased (Investigations) | 1
Insomnia (Psychiatric disorders) | 7
Intracranial hemorrhage (Nervous system disorders) | 1
Investigations - Other, specify (Investigations) | 1 — Elevated LDH
Lethargy (Nervous system disorders) | 1
Lung infection (Infections and infestations) | 6
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 1 — Iron deficiency anemia
Mucositis oral (Gastrointestinal disorders) | 1
Muscle cramp (Musculoskeletal and connective tissue disorders) | 1
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 — Muscle Aches
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1 — tendon rupture Left foot
Myalgia (Musculoskeletal and connective tissue disorders) | 5
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8
Nausea (Gastrointestinal disorders) | 18
Neck edema (General disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 3
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — nasal cavity mass
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — cyst
Neoplasms benign, malignant and unspecified (incl cysts and polyps) - Other, specify (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Basal cell carcinoma (Left upper arm and Left thigh)
Nervous system disorders - Other, specify (Nervous system disorders) | 2 — Neurotoxicity
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Lightheadedness
Nervous system disorders - Other, specify (Nervous system disorders) | 1 — Migraine
Neutrophil count decreased (Investigations) | 17
Non-cardiac chest pain (General disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 3
Pain (General disorders) | 13
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10
Pain of skin (Skin and subcutaneous tissue disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Papulopustular rash (Infections and infestations) | 2
Paresthesia (Nervous system disorders) | 2
Perineal pain (Reproductive system and breast disorders) | 1
Peripheral sensory neuropathy (Nervous system disorders) | 5
Platelet count decreased (Investigations) | 5
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Prostatic obstruction (Reproductive system and breast disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 4
Psychiatric disorders - Other, specify (Psychiatric disorders) | 1 — ADHD
Purpura (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Rectal pain (Gastrointestinal disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — Hydronephrosis
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — difficulty starting stream due to disease
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — BK Virus
Renal and urinary disorders - Other, specify (Renal and urinary disorders) | 1 — urinary hesitancy
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 1 — vaginal bleeding
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 — Chronic Obstructive Pulmonary Disease
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 2 — Asthma
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 1 — Seasonal Allergies
Seizure (Nervous system disorders) | 1
Sepsis (Infections and infestations) | 1
Sinus bradycardia (Cardiac disorders) | 1
Sinusitis (Infections and infestations) | 1
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Psoriasis to left foot
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Poison Ivy to Bilateral lower extremities and Left arm
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Rash, unspecified
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — growth on left cheek
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Skin tear - Right buttocks
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — weeping lesion
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — Fissure (coccyx)
Sinus tachycardia (Cardiac disorders) | 4
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 1 — multiple skin tears to Left and Right FA and Right heel
Skin infection (Infections and infestations) | 1
Skin ulceration (Skin and subcutaneous tissue disorders) | 2
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 2
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1
Somnolence (Nervous system disorders) | 1
Sore throat (Respiratory, thoracic and mediastinal disorders) | 6
Syncope (Nervous system disorders) | 1
Testosterone deficiency (Endocrine disorders) | 1
Thromboembolic event (Vascular disorders) | 3
Thrush (Infections and infestations) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Tremor (Nervous system disorders) | 6
Tumor lysis syndrome (Metabolism and nutrition disorders) | 1
Upper respiratory infection (Infections and infestations) | 3
Urinary frequency (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 6
Urinary retention (Renal and urinary disorders) | 3
Urinary tract infection (Infections and infestations) | 4
Urinary urgency (Renal and urinary disorders) | 1
Vaginal discharge (Reproductive system and breast disorders) | 1
Vaginal dryness (Reproductive system and breast disorders) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Ventricular tachycardia (Cardiac disorders) | 1
Vertigo (Ear and labyrinth disorders) | 1
Vomiting (Gastrointestinal disorders) | 6
Weight gain (Investigations) | 3
White blood cell decreased (Investigations) | 2
Weight loss (Investigations) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-06-10): https://cdn.clinicaltrials.gov/large-docs/49/NCT05583149/Prot_SAP_000.pdf